CLINICAL TRIAL: NCT00955812
Title: A Phase I, Open-label, Dose Escalation, Non-randomized Study to Assess the Pharmacokinetics, Dose Limiting Toxicity, and Maximum Tolerated Dose of OPB-31121 in Subjects With Advanced Solid Tumors
Brief Title: STAT3 Inhibitor for Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0206
Record Dates: First submitted 2009-08-07; First posted 2009-08-10 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Cancer; Solid Tumor
Keywords: OPB-31121; Advanced Solid Tumor; STAT3; IL-6-induced STAT3 phosphorylation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-31121 (Experimental): OPB-31121 50 mg by mouth 2 times a day on Days 1-21 of each 28-day cycle.
  Interventions: Drug: OPB-31121

INTERVENTIONS:
Drug: OPB-31121 — 50 mg by mouth 2 times a day on Days 1-21 of each 28-day cycle.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of OPB-31121 that can be given to patients with an advanced solid tumor. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

OPB-31121 is designed to block certain proteins in cancer cells that cause the cancer cells to reproduce and form more cancer cells.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of OPB-31121 based on when you joined this study. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of OPB-31121 is found.

Study Drug Administration:

On Days 1-21 of each 28-day cycle, you will take the study drug by mouth 2 times a day. You should take the study drug with at least 1 full glass of room temperature, still (non-carbonated) water, within 30 minutes after eating a snack or meal. You should either remain sitting upright or standing for at least 30 minutes after you take the study drug. You will be given directions by the study doctor, the study nurse, and/or the study pharmacist on how to take the study drug at home.

Study Visits:

On Day 1 of Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have 5 ECGs: 1 before the morning dose of study drug and at 1, 2, 4, and 8 hours after the morning dose.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 2 teaspoons each time) will be drawn before the morning dose and then 6 more times over the next 12 hours after the dose for pharmacokinetic (PK) testing. PK testing measures the amount of study drug in the body at different time points.
* Blood (about 2 teaspoons) for pharmacodynamic (PD) testing will be drawn before the morning dose. PD testing is used to look at how the level of study drug in your body may affect the disease.
* Blood (about 1 teaspoon) will be drawn for pharmacogenomic (PGx) testing. PGx testing looks at how differences in people's genes may affect if and how well the study drug may affect the disease.
* Women who are able to become pregnant will have a urine pregnancy test.

On Day 2 of Cycle 1, before your morning dose of study drug, the following tests and procedures will be performed:

* Blood (about 1 teaspoon) will be drawn for a troponin test.
* Blood (about 4 teaspoons) will be drawn for PK and PD testing.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.

On Days 8, 15, 21, and 28 of Cycle 1, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Blood (about 3 tablespoons on Days 8 and 15; about 1 tablespoon on Days 21 and 28) and urine will be collected for routine tests.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.

On Day 21 of Cycle 1, blood (about 2 teaspoons each time) will be drawn for PK testing before the morning dose and then 6 more times over the next 12 hours after the dose. Blood (about 2 teaspoons each time) will also be drawn for PD testing.

On Day 22 of Cycle 1, before your morning dose of study drug, the following tests and procedures will be performed:

* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.
* Blood (about 2 teaspoons) will be drawn for PK testing before your morning dose of the study drug.

On Days 1, 15, and 28 of Cycles 2 and beyond, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you had any side effects from them.
* You will have an ECG.
* You will have an echocardiogram or MUGA scan.
* Blood (about 3 tablespoons) will be drawn for routine tests.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Women who are able to become pregnant will have a urine pregnancy test.

About every 8 weeks, you will have an x-ray, CT scan, or MRI scan to check the status of the disease.

Length of Study:

You may continue taking the study drug for as long as you are benefitting. You will be taken off study if the disease gets worse, you experience intolerable side effects, or your doctor thinks that it is no longer in your best interest to receive the study drug.

You may choose to stop taking the study drug at any time. You should tell the study doctor right away if you are thinking about stopping your participation in this study. The study doctor will talk to you about how to safely stop taking the study drug.

End-of-Study Visi:t

Within 14 days after the last dose of study drug, you will return for a final visit. The following tests and procedures will be performed at the final visit:

* You will have a physical exam, including measurement of your vital signs.
* You will have an ECG.
* Blood (about 4 tablespoons) and urine will be collected for routine tests.
* You will have either an ECHO or MUGA scan.
* You will have an x-ray, CT scan, or MRI scan to check the status of the disease.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.

Follow-Up:

You will be called about 30 days after the last dose of OPB-31121 and asked if you have experienced any new or ongoing side effects.

This is an investigational study. OPB-31121 is not FDA approved or commercially available. At this time, OPB-31121 is only being used in research.

Up to 36 patients will take part in this multicenter study. Up to 18 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histologically or radiologically confirmed solid tumors refractory to standard therapy, for which there is no standard therapy, or are not eligible for standard therapy. Subjects must have at least one measurable lesion.
2. Male and female subjects >/= 18 years of age.
3. Male and female subjects who are surgically sterile; female subjects who have been postmenopausal for at least 12 consecutive months; or male and female subjects who agree to remain abstinent or to begin TWO acceptable methods of birth control from one week prior to drug administration through 30 days (for females) and 90 days (for males) from the last dose of study medication. If employing birth control, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device (IUD), condom, diaphragm, cervical cap or sponge with spermicide.
4. Eastern Cooperative Oncology Group (ECOG) performance status: </= 2
5. Subjects must have a life expectancy of longer than 3 months.
6. Adequate vital organ function as follows: Neutrophils: >/= 1,500/microliter; platelets: >/= 75,000/microliter; hemoglobin: >/= 9.0 g/dL; Aspartate transaminase (AST), Alanine transaminase (ALT): </= 2.5 * ULN with the exception of subjects with liver metastases. In these cases, AST, ALT </= 5 * ULN for eligibility; serum total bilirubin: < 2.5 * ULN. Subjects must have a normal serum creatinine with a measured 24 hour creatinine clearance of > 60 cc/min; INR < 1.5
7. Ability to provide written informed consent prior to initiation of any study-related procedures, and ability, in the opinion of the principal investigator, to comply with all the requirements of the study.
8. Subjects, who have received prior therapy, eg, chemotherapy, radiotherapy, or surgery, must have stopped therapy for >/= 4 weeks prior to drug administration. Subjects who have received targeted or immunotherapy must have stopped therapy for 5 half lives or 4 weeks prior to drug administration, whichever is earlier, and recovered from any prior toxicity not mentioned above to at least Grade 1.
9. Subjects must have a normal ejection fraction (>/= 50%) as measured by either echocardiogram or multi gated acquisition (MUGA) scan.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
2. Known central nervous system (CNS) metastasis.
3. Presence of active gastrointestinal disease or other condition (eg, significant bowel resections) which has the potential to significantly affect the absorption of the study drug, in the opinion of the investigator or sponsor.
4. Known history of or concurrent hepatitis or acquired immunodeficiency syndrome (AIDS) or known carriers of hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies (anti-HCV), or human immunodeficiency virus (HIV) antibodies.
5. Subjects who are pregnant or breast feeding. A negative urine pregnancy test must be confirmed prior to the first dose of study drug for women of child bearing potential (WOCBP).
6. Administration of another investigational agent within 28 days or 5 half-lives for targeted therapy or immunotherapy (whichever is shorter) prior to study entry
7. Use of prohibited medications
8. Subjects with history of coagulopathy (or taking anticoagulants) including deep vein thrombosis (DVT)/pulmonary embolism (PE), myocardial infarction or stroke within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of OPB-31121 | 4 Week Cycle
  The MTD is defined as the highest dose level at which < 2 of 6 subjects experience dose limiting toxicity (DLT) during the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Hong, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (2):
- United States (2):
  - Sarah Cannon Research Institute (SCRI), Nashville, Tennessee
  - UT MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Bendell JC, Hong DS, Burris HA 3rd, Naing A, Jones SF, Falchook G, Bricmont P, Elekes A, Rock EP, Kurzrock R. Phase 1, open-label, dose-escalation, and pharmacokinetic study of STAT3 inhibitor OPB-31121 in subjects with advanced solid tumors. Cancer Chemother Pharmacol. 2014 Jul;74(1):125-30. doi: 10.1007/s00280-014-2480-2. Epub 2014 May 13. PMID 24819685
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org